CLINICAL TRIAL: NCT05087836
Title: Correlation of Regional Cerebral Oxygen Saturation Monitoring by NIRS Between Standard Site vs Alternative Sites of Sensor Position in Adult Cardiac Surgery
Brief Title: Correlation of Cerebral Oxygen Saturation Measured From 2 Sensor Sites: Forehead vs. Temporal
Status: Completed | Type: Observational
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Thepakorn Sathitkarnmanee, Associate professor, Khon Kaen University
Other Study IDs: HE641311
Record Dates: First submitted 2021-10-09; First posted 2021-10-21 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Cerebral Ischemia
Keywords: NIRS; Regional cerebral oxygen saturation; sensor; forehead; temporal
MeSH Terms: conditions — Brain Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient undergoing cardiac surgery: Each patient will has 2 sets of sensors attached at forehead and temporal area.
  Interventions: Device: Sensor at forehead area; Device: Sensor at temporal area

INTERVENTIONS:
Device: Sensor at forehead area — NIRS sensor attached at forehead area.
Device: Sensor at temporal area — NIRS sensor attached at temporal area.

SUMMARY:
Cardiac surgery and neurosurgery may decrease cerebral blood flow leading to cerebral dysfunction. Regional cerebral oxygen saturation (rScO2) monitor via Near-infrared spectometry (NIRS) is recommended for early detection and correction. The standard site of NIRS sensor is forehead area which is impractical in operation with incision at forehead area. The investigators suggest an alternative sensor site at temporal area. The objective of this study is to assess the correlation of rScO2 measured from sensor attached at forehead vs. temporal area.

DETAILED DESCRIPTION:
Cardiac surgery and neurosurgery may decrease cerebral blood flow leading to neurologic morbidity, e.g., postoperative stroke, delirium, or postoperative cognitive dysfunction. Regional cerebral oxygen saturation (rScO2) monitor via Near-infrared spectometry (NIRS) is thus recommended for early detection and correction. Murkin et al.(2007) conducted a randomized controlled trial in coronary artery bypass graft (CABG) with NIRS monitoring showed that patients who received intervention to avoid rScO2 < 75% of baseline had less major organ morbidity including stroke, and mortality. Senanayake et al.(2012) revealed that NIRS could decrease neurologic complication in patients undergoing ascending aortic replacement with moderate hypothermic circulatory arrest.

The standard site of NIRS sensor is forehead area. There are some types of surgery involving incision at forehead area which makes it not possible to attach sensor at this site. The investigators propose an alternative sensor site at temporal area to be used in such situation.

The objective of this study is to assess the correlation of rScO2 measured from sensor attached at forehead vs. temporal area.

ELIGIBILITY:
Inclusion Criteria:

* age =/> 18 y
* undergoing elective cardiac surgery
* American Society of Anesthesiologists (ASA) classification II-III

Exclusion Criteria:

* history of intracranial or carotid vascular disease
* previous surgery at face or brain
* abnormal anatomy of face
* re-do surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
rScO2 | intraoperatively
  Regional cerebral oxygen saturation

CONTACTS AND LOCATIONS:
Overall Officials: Thepakorn Sathitkarnmanee, MD, Principal Investigator — Faculty of Medicine, Khon Kaen University, Khon kaen, Thailand
Locations (1):
- Faculty of Medicine, Khon Kaen University, Khon Kaen, Thailand

REFERENCES:
- [Result] Moerman A, Wouters P. Near-infrared spectroscopy (NIRS) monitoring in contemporary anesthesia and critical care. Acta Anaesthesiol Belg. 2010;61(4):185-94. PMID 21388077
- [Result] Murkin JM, Adams SJ, Novick RJ, Quantz M, Bainbridge D, Iglesias I, Cleland A, Schaefer B, Irwin B, Fox S. Monitoring brain oxygen saturation during coronary bypass surgery: a randomized, prospective study. Anesth Analg. 2007 Jan;104(1):51-8. doi: 10.1213/01.ane.0000246814.29362.f4. PMID 17179242
- [Result] Senanayake E, Komber M, Nassef A, Massey N, Cooper G. Effective cerebral protection using near-infrared spectroscopy monitoring with antegrade cerebral perfusion during aortic surgery. J Card Surg. 2012 Mar;27(2):211-6. doi: 10.1111/j.1540-8191.2012.01420.x. PMID 22458277
- [Result] Colak Z, Borojevic M, Bogovic A, Ivancan V, Biocina B, Majeric-Kogler V. Influence of intraoperative cerebral oximetry monitoring on neurocognitive function after coronary artery bypass surgery: a randomized, prospective study. Eur J Cardiothorac Surg. 2015 Mar;47(3):447-54. doi: 10.1093/ejcts/ezu193. Epub 2014 May 7. PMID 24810757
- [Result] Zheng F, Sheinberg R, Yee MS, Ono M, Zheng Y, Hogue CW. Cerebral near-infrared spectroscopy monitoring and neurologic outcomes in adult cardiac surgery patients: a systematic review. Anesth Analg. 2013 Mar;116(3):663-76. doi: 10.1213/ANE.0b013e318277a255. Epub 2012 Dec 24. PMID 23267000